CLINICAL TRIAL: NCT04683003
Title: A Phase 3b, Prospective, Open-label, Multicenter, Single Treatment Arm, Continuation Study of the Safety and Efficacy of TAK-755 (rADAMTS13, Also Known as BAX 930/SHP655) in the Prophylactic and On-demand Treatment of Subjects With Severe Congenital Thrombotic Thrombocytopenic Purpura (cTTP; Upshaw-Schulman Syndrome, or Hereditary Thrombotic Thrombocytopenic Purpura)
Brief Title: A Study of TAK-755 in Participants With Congenital Thrombotic Thrombocytopenic Purpura
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Collaborators: Takeda Development Center Americas, Inc. (Industry); Shire (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAK-755-3002; 2020-003348-10 (EudraCT Number)
Record Dates: First submitted 2020-12-10; First posted 2020-12-24 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Thrombotic Thrombocytopenic Purpura (TTP)
Keywords: Congenital Thrombotic Thrombocytopenic Purpura (TTP)
MeSH Terms: conditions — Purpura, Thrombotic Thrombocytopenic | interventions — ADAMTS13 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Prophylactic Cohort: TAK-755 (Experimental): All participants will receive prophylactic treatment with 40 IU/kg TAK-755 intravenous (IV) infusions once every week or once every other week for the duration of the study.
  Participants who are naïve will receive an initial IV dose of 40 IU/kg TAK-755 to allow measurement of the pharmacokinetics of TAK-755, followed by prophylactic treatment with 40 IU/kg TAK-755 by IV infusion once every week or once every other week for the duration of the study.
  Interventions: Biological: TAK-755
- On-Demand Cohort: TAK-755 (Experimental): Participants will receive daily IV infusions of TAK-755 when experiencing an acute thrombotic thrombocytopenic purpura (TTP) event until 2 days after the acute TTP event is resolved.
  Participants will receive 40 IU/kg TAK-755 on the first day, followed by 20 IU/kg on Day 2, and then 15 IU/kg daily until 2 days after the acute TTP event has resolved. Upon resolution of the acute TTP event, participants may choose to move to the prophylactic cohort of the study or discontinue entirely from the study.
  Interventions: Biological: TAK-755

INTERVENTIONS:
Biological: TAK-755 — TAK-755 IV infusion
  Other Names: rADAMTS13; recombinant ADAMTS13; SHP-655; BAX 930

SUMMARY:
Thrombotic thrombocytopenic purpura (or TTP for short) is a condition where blood clots form in small blood vessels throughout the body. The clots can limit or block the flow of oxygen-rich blood to the body's organs, such as the brain, kidneys, and heart. As a result, serious health problems can develop. The increased clotting that occurs in TTP uses up the cells that help the blood to clot, called platelets. With fewer platelets available in the blood, bleeding problems can also occur. People who have TTP may bleed underneath the skin forming purple bruises, or purpura. TTP also can cause anemia, a condition in which red blood cells break apart faster than the body can replace them, leading to fewer red blood cells than in normal.

TTP is caused by a lack of activity in the ADAMTS13 enzyme, a protein in the blood involved in controlling clotting of the blood. The ADAMTS13 enzyme breaks up another blood protein called von Willebrand factor that forms blood clots by clumping together with platelets. Some people are born with this condition, while others develop the condition during their life. Many people who are born with TTP experience frequent flare-ups that need to be treated right away. TAK-755 is a medicine that replaces ADAMTS13 and may prevent or control TTP flare-ups, called acute TTP events.

The main aim of the study is to check for side effects of long-term treatment with TAK-755. Treatment will be given in 2 ways:

1. TAK-755 treatment given either every week or every other week to prevent acute TTP events from happening (the "prophylactic" cohort).
2. TAK-755 treatment given to control an acute TTP event when it happens (the "on-demand" cohort).

Participants in the prophylactic cohort will receive treatment in the clinic or at home for up to approximately 3 years. They will visit the clinic at least every 12 weeks. Participants in the on-demand cohort will receive daily treatment for the acute TTP event until the flare-up has gotten better. They will have a follow-up visit at the clinic 4 weeks later.

DETAILED DESCRIPTION:
This is a follow-up study to the Phase 3 pivotal study (281102 [NCT03393975]) and will be comprised of two treatment cohorts (Prophylactic and On-demand) consisting of naïve and non-naïve participants who were born with TTP, with a total duration of approximately 6 years. A maximum of approximately 77 participants will be enrolled in this study (approximately 57 participants who have completed study 281102 [NCT03393975] [non-naïve participants] and at least 20 naïve participants (participants who are naïve to TAK-755). Participants from Expanded Access Programs, participants from study 281102 (NCT03393975) who had an allergic reaction to standard of care treatment, and participants who completed the Phase 1 study (281101 [NCT02216084]) but did not participate in Study 281102, will also be eligible for enrollment in this continuation study as naïve participants.

TAK-755 is given slowly through a vein (intravenous infusion). Participants in the prophylactic cohort will be able to opt for treatment in a home setting by caregiver or self-infusion subject to conditions and to local regulatory approval.

ELIGIBILITY:
Inclusion Criteria:

Participants who have completed TAK-755 Phase 3 pivotal Study 281102 (NCT03393975) in the prophylactic cohort and who meet all of the following criteria are eligible for this study:

* Participants or legally authorized representative has provided signed informed consent >=18 years of age and/or assent form <18 years of age.
* Participant 0 to 70 years of age at the time of screening of the 281102 (NCT03393975) study.
* Participant has been diagnosed with severe congenital ADAMTS-13 deficiency.
* Participant does not display any severe thrombotic thrombocytopenic purpura (TTP) signs (platelet count <100,000/ microliter (mcL) and elevation of lactate dehydrogenase (LDH) greater than (>) 2 × ULN at screening (prophylactic cohort only).
* Participants >=16 years of age must have a Karnofsky score >= 70% and participants <16 years of age must have a Lansky score >=80%.
* If female of childbearing potential, participant presents with a negative serum or urine pregnancy test confirmed not more than 7 days before the first IP administration and agrees to employ adequate birth control measures for the duration of the study and to undergo quarterly pregnancy testing.
* Sexually active males must use an accepted and effective method of contraception during the treatment and until a minimum of 16 days after the last dose administered.
* Participant is willing and able to comply with the requirements of the protocol.

All naïve participants and non-naïve on-demand cohort participants:

Naïve participants can only be enrolled in this continuation after enrollment of the adult participants in the prophylactic arm of TAK-755 Phase 3 pivotal study 281102 (NCT03393975) has been completed. Naïve pediatric participants can be enrolled after enrollment of the respective age cohort into the pivotal Phase 3 study 281102 (NCT03393975) has been completed. The following criteria also applies to participants who completed study 281101 (NCT02216084), but did not participate in 281102 (NCT03393975).

Naïve participants and participants who were enrolled into the on-demand cohort of theTAK-755 Phase 3 pivotal study 281102 (NCT03393975) who meet ALL of the following criteria are eligible for this study:

* Participant is naïve or was enrolled into the on-demand cohort of the TAK-755 Phase 3 pivotal study 281102 (NCT03393975) for treatment of an acute TTP event but did not receive prophylactic treatment.
* Participant or legally authorized representative has provided signed informed consent (>=18 years of age) and/or assent form (<18 years of age).
* Participant is 0 to 70 years of age at the time of screening.
* Participant has been diagnosed with severe congenital ADAMTS-13 deficiency defined as:

  * Confirmed by molecular genetic testing, documented in participant history or at screening, and
  * ADAMTS-13 activity <10% as measured by the fluorescence resonance energy transfer (FRETS)-VWF73 assay, documented in participant history or at screening. Participants currently receiving standard of care prophylactic therapy may exceed 10% ADAMTS-13 activity at screening.
* Participants currently receiving prophylactic therapy will be screened immediately prior to their usual prophylactic infusion.
* Participant does not display any severe TTP signs (platelet count <100,000/microliter (mcL) and elevation of LDH >2 × ULN) at screening (prophylactic cohort only).
* Participants >=16 years of age must have a Karnofsky score >=70% and participants <16 years of age must have a Lansky score >=80%.
* Participants is hepatitis C virus negative (HCV-) as confirmed by antibody or polymerase chain reaction testing OR HCV positive (HCV+) if their disease is chronic but stable.
* If female of childbearing potential, participant presents with a negative serum or urine pregnancy test confirmed not more than 7 days before the first IP administration and agrees to employ adequate birth control measures for the duration of the study and to undergo quarterly pregnancy testing.
* Sexually active males must use an accepted and effective method of contraception during treatment and until a minimum of 16 days after the last dose administered.
* Participant is willing and able to comply with the requirements of the protocol.

Participants from an Expanded Access Program or participants in Study 281102 (NCT03393975) who had an allergic reaction to standard of care prophylactic treatment must meet all of the following criteria:

Participants from an expanded access program as well as participants who participated in Study 281102(NCT03393975) who had an allergic reaction to standard-of-care prophylactic treatment are eligible for enrollment in the continuation study if they meet ALL of the following criteria.

* Participants or legally authorized representative has provided signed informed consent (>=18 years of age) and/or assent (<18 years of age).
* Participants is 0 to 70 years of age at the time of screening.
* Participants has been diagnosed with severe congenital ADAMTS-13 deficiency defined as:

  * Confirmed by molecular genetic testing, documented in participant history or at screening, and
  * ADAMTS-13 activity <10% as measured by the fluorescence resonance energy transfer (FRETS)- VWF 73 assay, documented in participant history or at screening. Participants currently receiving standard of care prophylactic therapy may exceed 10% ADAMTS 13 activity at screening.
* Participant does not display any severe TTP signs (platelet count <100,000/mcL and elevation of LDH >2 × ULN) at screening (prophylactic cohort only).
* Participants >=16 years of age must have a Karnofsky score >=70% and participants <16 years of age must have a Lansky score >=80%.
* If female of childbearing potential, participant presents with a negative serum or urine pregnancy test confirmed not more than 7 days before the first IP administration and agrees to employ highly effective birth control measures for the duration of the study and to undergo quarterly pregnancy testing.
* Sexually active males must use an accepted and effective method of contraception during treatment and until a minimum of 16 days after the last dose administered.
* Participant is willing and able to comply with the requirements of the protocol.

Exclusion Criteria:

Participants who have completed TAK-755 Phase 3 pivotal study (281102) (NCT03393975) and naïve participants and non-naïve on-demand cohort participants and participants from an Expanded Access Program or participants in Study 281102 (NCT03393975) who had an allergic reaction to standard-of-care prophylactic treatment. The following criteria also applies to participants who completed study 281101 (NCT02216084), but did not participate in 281102 (NCT03393975).

* Participant has been diagnosed with any other TTP-like disorder (microangiopathic hemolytic anemia), including immune-mediated TTP.
* Known life-threatening hypersensitivity reaction, including anaphylaxis, to the parent molecule ADAMTS-13, hamster protein, or other constituents of TAK-755.
* Participant has a presence of a functional ADAMTS-13 inhibitor at screening.
* Participant has a medical history of a genetic or acquired immune deficiency that would interfere with the assessment of product immunogenicity, including participants who are human immunodeficiency virus-positive with an absolute cluster of differentiation 4 (CD4) count < 200/ cubic millimeter (mm^3) or who are receiving chronic immunosuppressive drugs.
* Participant has a history of significant neurological events, such as major stroke, indicating that a relapse might have severe consequences, as judged by the investigator.
* Participant has been diagnosed with severe cardiovascular disease (New York Heart Association classes 3 to 4).
* Participant with end stage renal disease requiring chronic dialysis.
* Participant has been diagnosed with hepatic dysfunction, as evidenced by, but not limited to, any of the following:

  * Serum alanine aminotransferase >= 2 × ULN
  * Severe hypoalbuminemia <24 gram per liter (g/L)
  * Portal vein hypertension (e.g., presence of otherwise unexplained splenomegaly, history of esophageal varices).
* In the opinion of the investigator, the participant has another clinically significant concomitant disease that may pose additional risks for the participant.
* Participant has been treated with an immunomodulatory drug, excluding topical treatment (e.g., ointments, nasal sprays), within 30 days prior to enrollment. Use of corticosteroids in conjunction with administration of fresh frozen plasma to prevent allergic reactions is permitted.
* Participant has an acute illness (e.g., influenza, flu-like syndrome, allergic rhinitis/conjunctivitis, bronchial asthma) at the time of screening (prophylactic cohort only).
* Participant is receiving or anticipates receiving another investigational drug and/or interventional drug within 30 days before enrollment.
* Participant has a history of drug and/or alcohol abuse within the last 2 years.
* Participant has a progressive fatal disease and/or life expectancy of <= 3 months.
* Participant is identified by the investigator as being unable or unwilling to cooperate with study procedures.
* Participant suffers from a mental condition rendering him/her unable to understand the nature, scope, and possible consequences of the study and/or evidence of an uncooperative attitude.
* Participant is a family member or employee of the sponsor or investigator.
* If female, participant is pregnant or lactating at the time of enrollment.
* In the UK only: Participants who have not previously received a dose of TAK-755.

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 77 (Estimated)
Dates: Start 2021-04-14 (Actual); Primary Completion 2027-03-16 (Estimated); Study Completion 2027-03-16 (Estimated)

PRIMARY OUTCOMES:
Incidence of Related Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Throughout the study period of approximately 6 years
  TEAE: any adverse event emerging or manifesting at or after the initiation of treatment with TAK-755 or any existing adverse event that worsens in either intensity or frequency following exposure to TAK-755. SAE: Signs, symptoms or outcomes which results in death, requires inpatient hospitalization or prolongation of hospitalization, results in persistent or significant disability/incapacity, results in a congenital abnormality/birth defect, or is an important medical event.

SECONDARY OUTCOMES:
Number of Acute Thrombotic Thrombocytopenic Purpura (TTP) Events in Participants with Congenital Thrombotic Thrombocytopenic Purpura (cTTP) Undergoing Prophylactic Treatment with TAK-755 | Up to approximately 3 years
  The number of acute TTP Events in participants with cTTP receiving prophylactic treatment with TAK-755 (rADAMTS13) will be assessed.
Incidence Rate of Acute TTP Events in Participants with cTTP Undergoing Prophylactic Treatment with TAK-755 | Up to approximately 3 years
  Annualized acute TTP event incidence rate is calculated as the number of acute TTP events while receiving prophylactic treatment with TAK-755 (rADAMTS13) divided by the duration of the observation period in years. Annualized acute TTP event rate while participants are receiving prophylactic treatment with TAK-755 will be assessed.
Number of Acute TTP Events Resolved After Treatment with TAK-755 while Enrolled in the Study | Throughout the study period of approximately 6 years
  Acute TTP events are considered resolved when: Platelet count is >=150,000/ μL or platelet count is within 25% of baseline and elevation of lactate dehydrogenase (LDH) <= 1.5 x baseline or <= 1.5 x upper limit of normal (ULN).
Proportion of Acute TTP Events Resolved After Treatment with TAK-755 while Enrolled in the Study | Throughout the study period of approximately 6 years
  Proportion of acute TTP events that have resolved after treatment with TAK-755 (rADAMTS13) while enrolled in the study will be assessed. Acute TTP events are considered resolved when: Platelet count is >=150,000/ μL or platelet count is within 25% of baseline and elevation of LDH <= 1.5 x baseline or <= 1.5 x ULN.
Incidence of Acute TTP Events while Participants are on Their Final Dose and Dosing Regimen | Throughout the study period of approximately 6 years
  Incidence of annualized acute TTP events while participants are on their final dose and dosing regimen will be assessed.
Time to Resolution of Acute TTP Events Following Treatment with IP | Throughout the study period of approximately 6 years
  Time to resolution of acute TTP event is defined as the time from initial treatment of the event to resolution of the acute TTP event. Acute TTP events are considered resolved when: Platelet count is >=150,000/ μL or platelet count is within 25% of baseline and elevation of LDH <= 1.5 x baseline or <= 1.5 x ULN.
Total Quantity of TAK-755 Administered During the Treatment of Acute TTP Events | Throughout the study period of approximately 6 years
  Total quantity of TAK-755 administered during the treatment of acute TTP events will be assessed. Acute events typically require 3-4 days of intensified treatment.
Incidence of Supplemental Doses Prompted by Subacute TTP Events | Up to approximately 3 years
  Incidence of supplemental doses prompted by subacute TTP events in the prophylactic cohort will be assessed.
Incidence of Dose Modifications Not Prompted by an Acute TTP Event | Up to approximately 3 years
  Incidence of dose modifications not prompted by an acute TTP event in the prophylactic cohort will be assessed.
Incidence of Thrombocytopenia | Up to approximately 3 years
  Thrombocytopenia is defined as a drop in platelet count >=25 percent (%) of baseline or a platelet count less than (<) 150,000/mcL. Incidence of thrombocytopenia in the prophylactic cohort will be assessed.
Incidence of Microangiopathic Hemolytic Anemia | Up to approximately 3 years
  Microangiopathic hemolytic anemia is defined as an elevation of LDH greater than (>) 1.5xbaseline or LDH > 1.5xULN. Incidence of microangiopathic hemolytic anemia in the prophylactic cohort will be assessed.
Incidence of Neurological Symptoms | Up to approximately 3 years
  Neurological symptoms include headache, confusion, dysphonia, dysarthria, focal or general motor symptoms including seizures. Incidence of neurological symptoms in the prophylactic cohort will be assessed.
Incidence of Renal Dysfunction | Up to approximately 3 years
  Renal dysfunction is defined as an increase in serum creatinine >1.5xbaseline. Incidence of renal dysfunction in the prophylactic cohort will be assessed.
incidence of Abdominal Pain | Up to approximately 3 years
  Incidence of abdominal pain in the prophylactic cohort will be assessed.
Incidence of TTP Manifestations for Participants Receiving TAK-755 as a Prophylactic Treatment | Up to approximately 3 years
  TTP manifestations are defined as a composite of thrombocytopenia, microangiopathic hemolytic anemia, and TTP-related signs/symptoms including but not limited to (renal signs, neurologic symptoms, fever, fatigue/lethargy and abdominal pain). Incidence of TTP manifestations in the prophylactic cohort will be assessed.
Incidence of TTP Manifestations While Receiving the Final Prophylactic Treatment Regimen with TAK-755 in the Home Setting | Up to approximately 3 years
  TTP manifestations are defined as a composite of thrombocytopenia, microangiopathic hemolytic anemia, and TTP-related signs/symptoms including but not limited to (renal signs, neurologic symptoms, fever, fatigue/lethargy and abdominal pain). Incidence of TTP manifestations in the prophylactic cohort in the home setting will be assessed.
Incidence of Acute TTP Events in Participants Receiving TAK-755 Prophylactically in the Home Setting | Up to approximately 3 years
  Incidence of acute TTP events in participants receiving TAK-755 prophylactically in the home setting will be assessed.
Incidence of all AEs and SAEs (Including Unrelated) | Throughout the study period of approximately 6 years
  AE: any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this IP or medicinal product. SAE: Signs, symptoms or outcomes which results in death, requires inpatient hospitalization or prolongation of hospitalization, results in persistent or significant disability/incapacity, results in a congenital abnormality/birth defect, or is an important medical event.
Proportion of Participants with anti-ADAMTS13 Binding Antibodies and Neutralizing Antibodies Following ADAMTS13 Administration | Throughout the study period of approximately 6 years
  Proportion of participants with anti-ADAMTS13 binding antibodies and neutralizing antibodies following ADAMTS13 administration will be assessed.
Number of Participants Experiencing TAK-755 Related AEs and SAEs After Receiving TAK-755 in the Home Setting | Throughout the study period of approximately 6 years
  AE: Any untoward medical occurrence in a participant administered IP that does not necessarily have a causal relationship with the treatment. SAE: Signs, symptoms or outcomes which results in death, requires inpatient hospitalization or prolongation of hospitalization, results in persistent or significant disability/incapacity, results in a congenital abnormality/birth defect, or is an important medical event.
Number of Participants with AEs and SAEs After Receiving TAK-755 in the Home Setting | Throughout the study period of approximately 6 years
  AE: Any untoward medical occurrence in a participant administered IP that does not necessarily have a causal relationship with the treatment. SAE: Signs, symptoms or outcomes which results in death, requires inpatient hospitalization or prolongation of hospitalization, results in persistent or significant disability/incapacity, results in a congenital abnormality/birth defect, or is an important medical event.
Health Related Quality of Life (HRQoL): cTTP-Specific Patient reported outcomes (PROs) | Throughout the study period of approximately 6 years
  The cTTP specific patient-reported outcomes (PRO) instrument consists of 26 questions designed to assess the participants experience of fatigue, joint, muscle, abdominal and chest pain in the previous 24 hours, neurologic manifestations, bruising, feelings of depression and mood alterations, and activity limitation in the past 7 days, and participants attitudes, experienced side effects, work/school absences and travel impact associated with treatment received for TTP during the previous 2 weeks. The cTTP PRO assessment is focused on measuring the symptoms and impacts of the disease. The scores range from 0 to 152. Higher scores indicate a better quality of life.
HRQoL: 36-Item Short Form Health Survey (SF-36) | Throughout the study period of approximately 6 years
  The SF-36 is a generic quality-of-life instrument that has been widely used to assess HRQoL of participants. Generic instruments are used in general populations to assess a wide range of domains applicable to a variety of health states, conditions, and diseases. The SF-36 consists of 36 items that are aggregated into 8 multi-item scales (physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health), with scores ranging from 0 to 100. Higher scores indicate better HRQoL.
HRQoL: Abbreviated 9-item Treatment Satisfaction Questionnaire for Medication (TSQM-9) | Throughout the study period of approximately 6 years
  TSQM is a global satisfaction scale used to assess the overall level of participant's satisfaction or dissatisfaction with their medications. TSQM-9 is a 9-item, validated, self-administered instrument used to assess participant's satisfaction with medication. The three domains assessed are effectiveness, convenience, and global satisfaction. The score of each of the 3 domains is based on an algorithm to create a score of 0 to 100. Higher score indicated greater satisfaction in that domain.
HRQoL: EuroQol 5 Dimensions Questionnaire 3-Level (EQ-5D-3L) | Throughout the study period of approximately 6 years
  EQ-5D-3L health questionnaire is a participant answered questionnaire scoring 5 dimensions - mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The EQ-5D total score ranges from 0 (worst health state) to 1 (perfect health state) and 1 reflects the best outcome.
HRQoL: EQ-5D-youth (EQ-5D-Y) | Throughout the study period of approximately 6 years
  EQ-5D-Y health questionnaire is a participant answered questionnaire scoring 5 dimensions - mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The EQ-5D total score ranges from 0 (worst health state) to 1 (perfect health state) and 1 reflects the best outcome.
HRQoL: Pediatric Quality of Life Inventory (Peds QL) | Throughout the study period of approximately 6 years
  The Peds QL is a generic health related quality of life instrument designed specifically for a pediatric population and captures following domains: physical functioning, emotional functioning, social functioning, school functioning, psychosocial summary, physical health and total score. The Peds-QL total score consist of all 23 items of all domains. This modular instrument uses a 5-point scale: from 0 (never) to 4 (almost always). Items are reversed scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, 4=0. Higher scores indicate better quality of life.
HRQoL: Infusion Experience Satisfaction Assessment Questionnaire | Throughout the study period of approximately 6 years
  Infusion experience satisfaction assessment questionnaire will assess participant satisfaction on various aspects of the infusion experience (i.e., Convenience, impact on daily life, comfort in the treatment environment, time invested to receive infusion, concerns on handling potential complications, interaction with members of health care team and with other participants). Each item is rated on a 5-point scale from 1 (very poor) to 5 (very good) with a total score ranging from 93 to 465. Higher scores indicate greater satisfaction.
Resource Utilization: Length of Hospital Stay for Acute TTP Events | Throughout the study period of approximately 6 years
  Number of days of participants stay in hospital for acute TTP events will be assessed.
Resource Utilization: Number of Hospitalizations for Acute TTP Events | Throughout the study period of approximately 6 years
  Number of hospitalizations for acute TTP events will be assessed.
Resource Utilization: Number of Participants with Healthcare Resource Utilization During Prophylaxis | Up to approximately 3 years
  Health care resource utilization including days missed from school/work due to TTP-related illness will be assessed for the prophylactic cohort.
Resource Utilization: Number of Participants with Days Missed From School or Work due to TTP-Related Illness | Throughout the study period of approximately 6 years
  Number of participants with days missed from school or work due to TTP-related illness will be assessed.
Assessment of Trough and Postdose ADAMTS13 Activity: Antigen Levels (Activity:Ag) | At trough (for acute events) and within 72 hours pre-infusion and 65 minutes post-infusion (for both acute and subacute) at interval study visits every 12 weeks (up to 6 years)
  Trough and postdose ADAMTS13 activity and antigen levels from participants in prophylactic and on-demand cohorts during the study and during acute and subacute TTP events will be assessed.
Assessment of Von Willebrand Factor: Antigen (VWF:Ag) | At trough pre-infusion and 65 minutes post-infusion at interval study visits every 12 weeks (up to 6 years)
  VWF:Ag is a measure of total VWF protein and will be assessed using a sandwich enzyme-linked immunosorbent assay (ELISA) employing polyclonal anti-human-VWF antibodies. Assessments of VWF:Ag at baseline and following infusion of the TAK-755 treatment during the initial PK assessment in prophylactic and on-demand cohorts and during acute TTP events will be reported.
Assessment of Von Willebrand Factor: Ristocetin Cofactor Activity (VWF:RCo) | At trough pre-infusion and 65 minutes post-infusion at interval study visits every 12 weeks (up to 6 years)
  VWF:RCo will provide a measure of the ability of VWF to bind platelet glycoprotein Ib. Stabilized platelets are agglutinated in the presence of VWF and the antibiotic Ristocetin. Assessments of VWF:RCo during the study from participants in both the on-demand cohorts and during acute events will be reported.
Assessment of VWF:Ag in Relation to ADAMTS13 Activity Levels | At trough (for acute events) and within 72 hours pre-infusion and 65 minutes post-infusion (for both acute and subacute) at interval study visits every 12 weeks (up to 6 years)
  VWF:Ag is a measure of total VWF protein and will be assessed using a sandwich ELISA employing polyclonal anti-human-VWF antibodies. Longitudinal relationship of observed ADAMTS13 activity levels and VWF:Ag following infusion of the TAK-755 treatment during the initial PK assessment will be assessed (for TAK-755 naïve participants only).
Assessment of VWF:RCo in Relation to ADAMTS13 Activity Levels | At trough (for acute events) and within 72 hours pre-infusion and 65 minutes post-infusion (for both acute and subacute) at interval study visits every 12 weeks (up to 6 years)
  VWF:RCo will provide a measure of the ability of VWF to bind platelet glycoprotein Ib. Stabilized platelets are agglutinated in the presence of VWF and the antibiotic Ristocetin. Longitudinal relationship of observed ADAMTS13 activity levels and VWF:RCo following infusion of the TAK-755 treatment during the initial PK assessment will be assessed (for TAK-755 naïve participants only).
Number of Participants with Acute and Subacute Events in Relation with ADAMTS13 Activity Levels | At trough (for acute events) and within 72 hours pre-infusion and 65 minutes post-infusion (for both acute and subacute) at interval study visits every 12 weeks (up to 6 years)
  Longitudinal relationship of ADAMTS13 activity levels and participants with acute and subacute TTP events will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (27):
- United States (5):
  - Childrens Healthcare of Atlanta, Atlanta, Georgia
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Duke University Medical Center, Durham, North Carolina
  - Mid Ohio Heart Clinic Inc, Dublin, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
- AKH - Medizinische Universität Wien, Vienna, Austria
- China (5):
  - Beijing Children's Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Tongji Hospital Affiliated to Tongji Medicine University, Wuhan, Hubei
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsushe
  - Institute of Hematology and Hospital of Blood Disease, Tianjin, Tianjin Municipality
- France (4):
  - Hôpital Necker - Enfants Malades, Paris, Paris
  - CHU Saint Etienne - Hôpital Nord, Saint-Priest-en-Jarez Cedex, Pays de la Loire Region
  - Hôpital Saint-Antoine, Paris
  - Hôpital Robert Debré- Paris, Paris
- Germany (2):
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Universitaetsklinikum Jena, Klinik fuerKinder-und Jugendmedizin, Jena
- Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII (Presidio Papa Giovanni XXIII), Bergamo, Hubei, Italy
- Japan (3):
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Hyogo College of Medicine Hospital, Nishinomiya, Hyōgo
  - Medical Hospital,Tokyo Medical and Dental University, Bunkyo City, Tokyo
- Poland (2):
  - Samodzielny Publiczny Dzieciecy Szpital Kliniczny, Warsaw
  - Instytut Hematologii i Transfuzjologii, Warsaw
- Spain (2):
  - Complejo Hospitalario Universitario A Coruña, A Coruña, La Coruña
  - Hospital de Cruces, Barakaldo, Vizcaya
- Inselspital -Universitaetsspital Bern, Bern, Switzerland
- University College London Hospitals, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link. — https://clinicaltrials.takeda.com/study-detail/609976821f1122001e30a776?idFilter=%5B%22TAK-755-3002%22%5D